CLINICAL TRIAL: NCT05797389
Title: Effects of Graft Vascular Dimensions on Perioperative Surgical and Functional Outcomes of Living Donor Kidney Transplantation in Pediatrics and Adults: A Prospective Case Series
Brief Title: Effects of Graft Vascular Dimensions on Surgical and Functional Outcomes of Living Donor Kidney Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Loay, Assistant lecturer, Assiut University
Other Study IDs: vascular dimensions and KT
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Kidney Transplant; Complications
Keywords: kidney transplantation; renal transplantation; vascular dimensions; vascular parameters

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Correlate the radiological and intraoperative measuring of the vascular dimensions,
2. Assess the effect of the vascular dimensions on the short-term surgical complications and
3. Assess the effect of the vascular dimensions on the primary graft function in pediatric and adults KTs.

DETAILED DESCRIPTION:
Vascular complications after kidney transplantation (KT) are variably rare with an incidence of 3-15%. They are a significant and most serious part of surgical complications of KT. They may acutely result in graft loss during surgery or early in the perioperative period and may threaten patient's life. The most common forms of early vascular complications are haemorrhage, hematomas, arterial or venous thrombosis, arterial vasospasm, and arterial intimal dissection. In pediatric and adult KT, most studies addressing the vascular complications followed a common attitude of estimating the prevalence and management of these complications rather than studying the predisposing factors. Specifically, studying the normal and abnormal anatomy of the grafts has mainly been directed towards the number of graft vessels. However, there are many other vascular parameters that may potentially influence the outcome of vascular anastomosis and therefore the graft and patient outcomes. To the best of the investigators knowledge, the vascular dimensions of the renal and iliac vessels, such as the length, diameter and site of anastomosis to the iliac vessels have not been studied before so the investigators hypothesis that these dimensions can unequally affect the outcomes of surgery and early graft function in KTs. Hence, this study will be conducted to assess the effects of the vascular dimensions on the outcomes of surgery and primary graft function in pediatric versus adult living donor KT.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and adult patients undergoing living donor kidney transplantation.

Exclusion Criteria:

* Patients with acute graft rejection occurring within the first week of transplantation.
* Patients refusing participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult patients undergoing living donor kidney transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Mode of graft function defined by: 1- the time of start of diuresis post-transplantation. | one month post operative.
  Mode of graft function defined by:
  1- the start of diuresis (sufficient amount of urine production) within one hour of declamping through the first week post-transplantation
2- Rate of decline of the serum creatinine level. | one month post operative.
  2- Rate of decline of the serum creatinine level.

SECONDARY OUTCOMES:
The rate of vascular complications (intra- or perioperative). | one month post operative
  The rate of vascular complications (intra- or perioperative): In the form of spasm, hemorrhage, dissection, or thrombosis.
The rate of other surgical complications. | one month post operative
  The rate of other surgical complications.

REFERENCES:
- [Background] Srivastava A, Kumar J, Sharma S, Abhishek, Ansari MS, Kapoor R. Vascular complication in live related renal transplant: An experience of 1945 cases. Indian J Urol. 2013 Jan;29(1):42-7. doi: 10.4103/0970-1591.109983. PMID 23671364
- [Background] Fananapazir G, Troppmann C. Vascular complications in kidney transplant recipients. Abdom Radiol (NY). 2018 Oct;43(10):2546-2554. doi: 10.1007/s00261-018-1529-9. PMID 29500646
- [Background] Dimitroulis D, Bokos J, Zavos G, Nikiteas N, Karidis NP, Katsaronis P, Kostakis A. Vascular complications in renal transplantation: a single-center experience in 1367 renal transplantations and review of the literature. Transplant Proc. 2009 Jun;41(5):1609-14. doi: 10.1016/j.transproceed.2009.02.077. PMID 19545690
- [Background] Kadakia Y, Hwang C, MacConmara M. Rescue of an asymptomatic arterial occlusion after kidney transplant. BMJ Case Rep. 2022 Feb 7;15(2):e247347. doi: 10.1136/bcr-2021-247347. PMID 35131794
- [Background] Meltzer AZ, Fintha A, Cseprekal O, Somogyi D, Szabo J, Kobori L, Rozsa B, Piros L, Huszty G. Graft Arterial Dissection and Thrombosis After Kidney Transplantation With Undiagnosed Fibromuscular Dysplasia From a Deceased Donor: Case Report and Review. Transplant Proc. 2022 Nov;54(9):2603-2607. doi: 10.1016/j.transproceed.2022.10.049. Epub 2022 Nov 16. PMID 36400588
- [Background] Singh D, Butala BP, Parikh GP. Acute renal artery spasm during live kidney transplant surgery due to iatrogenic cause. Saudi J Kidney Dis Transpl. 2016 Mar;27(2):415-6. doi: 10.4103/1319-2442.178588. No abstract available. PMID 26997403
- [Background] Sevmis M, Demir ME, Merhametsiz O, Aktas S, Sevmis S, Uyar M. Grafts With Multiple Renal Arteries in Kidney Transplantation. Transplant Proc. 2021 Apr;53(3):933-940. doi: 10.1016/j.transproceed.2020.07.019. Epub 2020 Sep 17. PMID 32950261
- [Background] Ali-El-Dein B, Osman Y, Shokeir AA, Shehab El-Dein AB, Sheashaa H, Ghoneim MA. Multiple arteries in live donor renal transplantation: surgical aspects and outcomes. J Urol. 2003 Jun;169(6):2013-7. doi: 10.1097/01.ju.0000067637.83503.3e. PMID 12771707
- [Background] Osman Y, Shokeir A, Ali-el-Dein B, Tantawy M, Wafa EW, el-Dein AB, Ghoneim MA. Vascular complications after live donor renal transplantation: study of risk factors and effects on graft and patient survival. J Urol. 2003 Mar;169(3):859-62. doi: 10.1097/01.ju.0000050225.74647.5a. PMID 12576799
- [Background] Riella J, Tabbara MM, Alvarez A, DeFreitas MJ, Chandar J, Gaynor JJ, Gonzalez J, Ciancio G. Pediatric kidney transplants with multiple renal arteries show no increased risk of complications compared to single renal artery grafts. Front Pediatr. 2022 Dec 16;10:1058823. doi: 10.3389/fped.2022.1058823. eCollection 2022. PMID 36589161